CLINICAL TRIAL: NCT05953545
Title: Open Label Phase 2 Clinical Study of Peginterferon Lambda and Lonafarnib Boosted With Ritonavir 48-Week Combination Therapy for Delta Hepatitis
Brief Title: Peginterferon Lambda and Lonafarnib Boosted With Ritonavir 48-Week Combination Therapy for Delta Hepatitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closure based on decision of the PI
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001515; 001515-DK
Record Dates: First submitted 2023-07-19; First posted 2023-07-20 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Chronic Hepatitis Delta
Keywords: Hepatitis D; pegylated interferon lambda; Sustained Virological Response
MeSH Terms: conditions — Hepatitis D, Chronic; Hepatitis D | interventions — peginterferon lambda-1a

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Peginterferon Lambda (Experimental): A weekly subcutaneous injection of peginterferon lambda at a dose of 180 mcg and an oral twice daily dosing of Lonafarnib at 50mg boosted with twice daily Ritonavir at 100mg for 48 weeks. Following 48 weeks of treatment the subjects will be monitored for outcomes during an additional 6-month time period.
  Interventions: Drug: Peginterferon Lambda

INTERVENTIONS:
Drug: Peginterferon Lambda — Study intervention for this protocol includes a weekly subcutaneous injection of peginterferon lambda at a dose of 180 mcg and an oral twice daily dosing of Lonafarnib at 50mg boosted with twice daily Ritonavir at 100mg for 48 weeks. Following 48 weeks of treatment the subjects will be monitored for outcomes during an additional 6-month time period.

SUMMARY:
Background:

Chronic hepatitis D is a serious liver disease caused by a virus. Currently, no medications are approved to treat chronic hepatitis D.

Objective:

To test a combination of 3 drugs in people with chronic hepatitis D.

Eligibility:

People 18 years or older with chronic hepatitis D.

Design:

Participants will be in the study about 2 years. They will have 3 inpatient stays of 3 to 5 days.

Participants will be screened. They will have a physical exam with blood tests. They will have a test of their heart function and an ultrasound: a wand that uses sound waves to create images of the liver will be rubbed over the skin on their torso.

Participants will stay in the clinic for a 3-day baseline visit. They will have imaging scans, an eye exam, and a visit with a reproductive specialist. They will have a liver biopsy: about 1 inch of liver tissue will be removed, either with a tube inserted through a vein in the neck, or with a needle inserted through the participant s side.

Participants will take the study drugs for 48 weeks. Two of them are tablets taken twice a day at home; 1 is a shot administered once a week. Participants will begin taking the drugs during a 5-day stay in the clinic. Then they will have 15 outpatient visits while taking the drugs and 7 more after they finish.

The last 3-day clinic stay will be 6 months after participants finish taking the drugs. The liver biopsy, imaging scans, and other tests will be repeated.

DETAILED DESCRIPTION:
Study Description:

This is an open-label clinical trial treating 30 adult patients with chronic delta hepatitis with peginterferon lambda and lonafarnib boosted with ritonavir for 48 weeks. This is a follow up study to the previous 24-week combination study we had previously completed which demonstrated promising results. We hypothesize that therapy with peginterferon lambda and lonafarnib boosted with ritonavir will lead to a significant decline in hepatitis D virus RNA levels.

Objectives:

Primary Objective:

The goal of this study is to assess the therapeutic response to 48 weeks of treatment with peginterferon lambda and lonafarnib boosted with ritonavir in patients with chronic hepatitis D.

Secondary Objectives:

* Evaluation of the hepatitis D viral response to treatment during the treatment period and 24 weeks after the end of study.
* Evaluation of the hepatitis B viral response to treatment during the treatment period and 24 weeks after the end of study.
* Comparison of the patients liver parenchyma before and after treatment.
* Comparison of the patients liver biochemistry before, during and after treatment.
* Comparison of the patients hepatic venous pressure measurements before and after treatment.
* Evaluation of the patients bone density changes during therapy.
* Evaluation of changes in the patients fecal microbiome before, during and after treatment.
* Evaluation of the patients quality of life before, during and after treatment.

Tertiary Objective:

1. Comparison of the patients immune response before, during and after treatment.

Endpoints:

Primary Endpoint:

* Number of patients with HDV RNA levels < Lower Limit of Quantification (LLOQ), target not detected (TND) and the number of patients with HDV RNA levels <LLOQ, target detected (TD) in serum at 24 weeks after a 48-week treatment course of Peginterferon Lambda and Lonafarnib boosted Ritonavir.
* The ability to tolerate peginterferon lambda and lonafarnib boosted with ritonavir therapy for 48 weeks. Discontinuation of the medication by the clinical team or patient will be considered a failure to tolerate the medicine.

Secondary Endpoints:

* Sustained undetectable HDV RNA in serum at 48 weeks of treatment.
* Decrease of HDV RNA by >2 log from baseline at 48 weeks of therapy and 24 weeks post treatment.
* Determine the proportion of subjects with serum HDV RNA<LLOQ, TND with ALT normalization and <LLOQ, TD with ALT normalization.
* Reduction in histologic inflammatory scores (modified HAI) by at least two points with no progression in histologic fibrosis (Ishak) at week 24 post-treatment follow-up.
* Normalization of serum ALT (per reference lab) at the end of therapy and at week 24 of post-therapy follow-up, OR reduction in serum ALT by >50% of baseline at the end of therapy and week 24 of post therapy follow up.
* Reduction in hepatic venous pressure gradient (HVPG) measurements by >25% of baseline OR normalization of HVPG (<5 mm Hg) at week 24 post-treatment measurement.
* Reduction in Fibroscan(R) transient elastography values by >25% of baseline at study end.
* Loss of HBsAg from the serum at the end of therapy or at week 24 of post-therapy follow-up.
* Changes in quantitative HBsAg levels at the end of therapy and at week 24 of post therapy follow up, compared to baseline.
* Changes in bone density measurements by Dual-Energy X-ray Absorptiometry (DEXA).
* Changes in symptom scale measurements and quality of life before, during and after therapy.
* Changes in the fecal microbiome before, during and after treatment.

Tertiary endpoint:

-Changes in the patients peripheral blood mononuclear cell (PBMC) response to HDV during and following therapy in comparison to baseline. Changes in the phenotype and transcriptome of the intrahepatic immune cell infiltrate prior to and 24 weeks post end of therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Male or female, >=18 years of age.
* Presence of HDV RNA in serum at two points at least one day apart with HDV RNA levels that are quantifiable and above the lower limit of quantification (LLOQ) of the HDV RNA assay.
* Ongoing use of either tenofovir (TDF or TAF) or Entecavir for viral suppression of HBV for at least 12 weeks with documented suppression of HBV DNA (<100 IU/ml).

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Decompensated liver disease, defined by either bilirubin >2mg/dL, albumin <3.0 gm/dL, prothrombin time >2 sec prolonged, or history of bleeding esophageal varices, ascites, or hepatic encephalopathy. Laboratory abnormalities that are not thought to be due to liver disease may not necessarily require exclusion. Patients with an absolute neutrophil count <1000/dL and platelets <75,000/dL will be excluded from the study as well.
* Pregnancy or lactation.
* For females of reproductive potential: Lack of use of highly effective contraception defined as tubal ligation in women, or use of two contraceptive methods such as condoms (male partner) and spermicide in combination with an intrauterine device or a progestin-based hormonal contraception (implant or injection) for at least 3 months prior to treatment until 24 weeks after end of study medication administration. Female participants with childbearing potential must not use oral birth control pills as a form of contraception due to concern for interaction with study medications leading to contraception failure.
* For males of reproductive potential: Unable or unwilling to use condoms consistently in addition to female partner using another adequate contraceptive method to ensure effective contraception with partner during study participation and for an additional 24 weeks after the end of study medication administration. Patients who have undergone surgical sterilization (vasectomy) will still require female partner to utilize an additional adequate contraception method.
* Inability to take oral and subcutaneous medications
* Unwilling to adhere to the study intervention regimen or to comply with study procedures, or unavailability for the duration of the study
* Significant systemic or major illnesses other than liver disease, including, but not limited to, congestive heart failure, renal failure (eGFR <50 ml/min), organ transplantation, serious psychiatric disease or depression (only if felt to be at high risk by the NIH psychiatric consultation service), or active coronary artery disease.
* Systemic immunosuppressive therapy within the previous 2 months before enrollment.
* Evidence of another form of liver disease in addition to viral hepatitis (for example autoimmune liver disease, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson disease, alcoholic liver disease, ongoing drug induced liver disease, nonalcoholic steatohepatitis (but not steatosis), hemochromatosis, or alpha-1-antitrypsin deficiency).
* Active substance abuse, such as alcohol, inhaled or injection drugs within the previous year as determined by self-report or previous medical records.
* Evidence of hepatocellular carcinoma. This will be determined on the basis of imaging with ultrasound/ CT scan or MRI performed a maximum of 6 months prior to enrollment. Elevated AFP levels will be evaluated clinically, and further imaging may be performed if felt necessary.
* Evidence of concurrent hepatitis C infection with positive serum HCV RNA.
* Any experimental therapy, previous use of lonafarnib or pegylated interferon therapy within 6 months prior to enrollment.
* Active, serious autoimmune disease such as systemic lupus erythematosus, ulcerative colitis, Crohn s disease or rheumatoid arthritis, that is in the opinion of the investigators might be exacerbated by therapy with lambda interferon. This will be evaluated at baseline and during follow-up laboratory testing (including blood and urine studies) in addition to described symptoms at each outpatient visit.
* Diagnosis of malignancy in the five years prior to the enrollment with exception granted to superficial dermatologic malignancies.
* Evidence of HIV co-infection; HIV 1/2 antibody positivity on serum testing.
* Concurrent usage of statins as these drugs inhibits mevalonate synthesis, which reduces protein prenylation.
* Concurrent usage of moderate and strong CYP3A inhibitors and inducers.
* Concurrent usage of alpha 1 adrenoreceptor antagonist, antiarrhythmic, pimozide, sildenafil, sedative and hypnotics, ergot and St. John s Wort due to possible effect of ritonavir on hepatic metabolism of these drugs resulting in potentially life-threatening side effects.
* Clinically significant baseline EKG abnormalities such as QTc interval >450 ms and/or prolonged PR interval.
* Uncontrolled elevated triglycerides (>500 mg/dL). Patients on lipid lowering therapy other than statins will be eligible for this study.
* History of pancreatitis from causes other than gallstone pancreatitis. Subjects with a baseline amylase and/or lipase level >3 ULN will be excluded from the study.
* Any other condition, which in the opinion of the investigators would impede the patient s participation or compliance in the study.
* Inability to provide written informed consent.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
The goal of this study is to assess the therapeutic response to 48 weeks of treatment with peginterferon lambda and lonafarnib boosted with ritonavir in patients with chronic hepatitis D. | 48 weeks
  This is a phase 2 study evaluating the efficacy and safety of a novel regimen for the treatment of chronic HDV infection.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Koh, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001515-DK.html